CLINICAL TRIAL: NCT04359732
Title: Prediction of Assessment of Response to Neoadjuvant Chemo-Radio-Therapy (nCRT) for Esophageal and Gastroesophageal Junction Cancer (GEJ) Using a Fully Integrated PET/MRI
Brief Title: Assessment of Response to nCRT for GEJ Cancer Using a Fully Integrated PET/MRI
Acronym: Escape
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Principal Investigator, Francesco De Cobelli, MD, Chair Radiology Department, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Escape
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Cancer; Esophageal Neoplasms
Keywords: response; neoadjuvant; PET/MRI; radiomics; GEJ cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid PET/MRI (Other): For the purposes of the study, in addition to standard imaging (EUS and CT scan), a fully integrated hybrid PET/MRI (PET/MRI) study with FDG will replace the Standard PET (pre-surgical evaluation) used for evaluating distant metastases and will be considered as the add-on procedure at three time points. The additional evaluation for patients is that during nCRT treatment.
  Interventions: Other: hybrid PET/MRI

INTERVENTIONS:
Other: hybrid PET/MRI — An additional intermediate 18-FDG PET/MRI will be performed during neoadjuvant chemo-radiation therapy. Routine pre-treatment work-up PET/MRI will replace PET alone.

SUMMARY:
Evaluate the potential role of PET/MRI as a predictor of esophageal and junctional cancers in response to neoadjuvant chemoradiotherapy (nCRT).

DETAILED DESCRIPTION:
This is a prospective, observational single center study which plans to enroll patients with biopsy proven potentially resectable esophageal or junctional cancer scheduled to receive nCRT (CROSS regimen) prior to surgery.

The study aims to evaluate Routine pre-treatment work-up includes PET to stage the tumour extension.

* PET/MRI (Magnetic resonance imaging) will replace the PET component of CT(computed tomography)
* An additional intermediate 18-FDG (Fluorodeoxyglucose) PET/MRI will be performed during nCRT
* Post nCRT imaging, as required prior to surgery, will be PET/MRI six weeks after treatment completion.
* 8-12 weeks post nCRT completion surgery will be performed, based on each patient's performance status and response to nCRT
* Histopathological samples of the excised tumor and lymph nodes will be used for diagnosis, staging and description of qualitative and quantitative parameters Routine clinical and radiological follow-up for 24 months (for the scope of this study) will follow the standard clinical workflow assigned to this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven esophageal or junctional carcinomas (either adenocarcinoma (AC) or squamous cell carcinoma (SCC) for which an Ivor-Lewis transthoracic esophagectomy with supramesocolic and mediastinal lymphadenectomy is indicated;
* visible tumor on pre-treatment imaging;
* ≥ 18 years of age;
* signed informed consent.

Exclusion Criteria:

* - incomplete preoperative imaging assessment;
* contraindications to neoadjuvant treatment;
* contraindications to preoperative imaging (such as pacemaker, allergy to contrast agents);
* inability to complete imaging examinations (i.e. severe claustrophobia);
* contraindication to surgery (comorbidities, distant metastatic disease (imaging confirmed));
* pregnant or lactating women
* severe hypersensitivity to gadobutrol or fludeoxyglucose F18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Response to neoadjuvant treatment -MRI | 0-36 months
  MRI component including Dynamic Contrast Enhanced (DCE); quantitative evaluation and delta between timepoints
Response to neoadjuvant treatment -PET | 0-36 months
  PET component -quantitative evaluation and delta between timepoints
Response to neoadjuvant treatment - Histology | 0-36 months
  Evaluate degree of tumor regression after neoadjuvant therapy according to the Mandard Tumour regression grade ; integrated Immunohistochemistry
Response to neoadjuvant treatment -Radiomics | 0-36 months
  Radiomic features extracted from hybrid imaging
Imaging parameters as potential predictors of tumor response | 0- 48 months
  Select imaging parameters that can be considered potential predictors of the responder/non-responder status assessment

SECONDARY OUTCOMES:
Early regression model (ERI) | 0- 60 months
  Evaluate the ERI model as a predictor of histological response (TRG grade) based on MRI tumor volume assessment

CONTACTS AND LOCATIONS:
Overall Officials: Francesco De Cobelli, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Deaprtment of Radiology, IRCCS Ospedale San Raffaele, Milan, Italy